CLINICAL TRIAL: NCT00433173
Title: Effect of Increasing Testosterone on Insulin Sensitivity in Men With the Metabolic Syndrome
Brief Title: Insulin Sensitivity in Men With the Metabolic Syndrome
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary investigator is taking a leave of absence
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: American Diabetes Association (Other)
Responsible Party: Frances J. Hayes, MD, Massachusetts General Hospital, Boston MA 02114
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DK71168 (suspended); NIDDK # 1 RO1 DK071168-01A2
Record Dates: First submitted 2007-02-08; First posted 2007-02-09 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Metabolic Syndrome
Keywords: testosterone; insulin sensitivity; insulin resistance; metabolic disorders
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Metabolic Diseases | interventions — Glucose Tolerance Test; Testosterone; Anastrozole; Goserelin; Energy Metabolism; Absorptiometry, Photon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): 1) Group 1: Placebo
  Interventions: Procedure: intravenous glucose tolerance test; Procedure: aerobic capacity (VO2 Max); Procedure: MRI; Procedure: muscle biopsy; Procedure: measurement of resting metabolic rate (energy expenditure); Procedure: Dual energy x-ray absorptiometry; Procedure: Fasting oral glucose tolerance test
- 2 (Active Comparator): 2) Group 2: Depot GnRH agonist (Zoladex) + Testosterone + placebo
  Interventions: Procedure: intravenous glucose tolerance test; Drug: testosterone; Drug: goserelin acetate implant; Procedure: aerobic capacity (VO2 Max); Procedure: MRI; Procedure: muscle biopsy; Procedure: measurement of resting metabolic rate (energy expenditure); Procedure: Dual energy x-ray absorptiometry; Procedure: Fasting oral glucose tolerance test
- 3 (Active Comparator): 3) Group 3: (Zoladex + Testosterone + aromatase inhibitor (anastrozole)
  Interventions: Procedure: intravenous glucose tolerance test; Drug: testosterone; Drug: anastrozole; Drug: goserelin acetate implant; Procedure: aerobic capacity (VO2 Max); Procedure: MRI; Procedure: muscle biopsy; Procedure: measurement of resting metabolic rate (energy expenditure); Procedure: Dual energy x-ray absorptiometry; Procedure: Fasting oral glucose tolerance test

INTERVENTIONS:
Procedure: intravenous glucose tolerance test — The IVGTT (70) is a 4 hour study with baseline sampling for insulin and glucose, followed by the administration of 0.3 mg/kg infusion of glucose, and subsequent frequent samples through 180 minutes. At 20 minutes, subjects will receive a 0.03 U/kg infusion of regular human insulin over 45 seconds to enhance the insulin level to better help us assess the impact of insulin on glucose uptake and to facilitate minimal model analysis. The IVGTT will be administered at baseline and after 3 months.
  Other Names: IVGTT
Drug: testosterone — transdermal 7.5 g/per day for 3 months
  Other Names: Androgel 1%
  Arms: 2; 3
Drug: anastrozole — tablet (per oral) 10.0 mg/ daily 3 months
  Other Names: arimidex; IND# 76,878
  Arms: 3
Drug: goserelin acetate implant — single depot injection 10.8 mg 3 months
  Other Names: Zoladex
  Arms: 2; 3
Procedure: aerobic capacity (VO2 Max) — This test is employed to assess VO2max in all subjects. O2 and CO2 will be collected and measured from the expired air during the exercise stress test and used to calculate VO2max. This test will be administered at baseline and after 3 months.
Procedure: MRI — 1H-MR spectroscopy will be performed to measure IMCL at baseline and after 3 months.
Procedure: muscle biopsy — Biopsies (20-50mg) will be obtained from the vastus lateralis muscle under local anesthesia (1% lidocaine) using a 5 mm Bergström needle (65) with suction applied. The muscle biopsy will be performed at baseline and after 3 months.
Procedure: measurement of resting metabolic rate (energy expenditure) — Energy expenditure in the form of resting metabolic rate (RMR) will be measured via a metabolic monitor at baseline and after 3 months.
Procedure: Dual energy x-ray absorptiometry — Total and regional percent body fat, fat mass, lean tissue mass and bone mineral content will be determined by DEXA (Lunar Prodigy version 8.50). DEXA provides an in vivo assessment of body composition with minimal requirements for subject cooperation and will be employed at baseline and after 3 months.
  Other Names: DEXA
Procedure: Fasting oral glucose tolerance test — To examine glucose and insulin metabolism a standard 75g OGTT will be conducted at baseline and after 3 months.
  Other Names: OGTT

SUMMARY:
The metabolic syndrome is a medical condition defined by high levels of cholesterol in the blood, high blood pressure, central obesity (gain in fat around the region of the stomach), and insulin resistance (body responds less well to insulin). This state of impaired insulin resistance can lead to type 2 diabetes mellitus, which is one of the most common metabolic disorders in the U.S. Numerous studies have shown an inverse relationship between insulin resistance and testosterone levels in men, however, causality has not been established. This protocol investigates the role of testosterone in modulating insulin sensitivity in insulin resistant states such as the metabolic syndrome. The hypothesis is that testosterone administration will improve insulin sensitivity.

DETAILED DESCRIPTION:
This protocol will address the impact of three months of testosterone (T) therapy on all components of the metabolic syndrome and the mechanism underlying changes in insulin sensitivity by analyzing changes in body composition, and detailed studies of fat metabolism and skeletal muscle. In addition, this protocol will address the role of estradiol (E2) in mediating the effect of testosterone on insulin sensitivity.

Seventy-two subjects will be enrolled. Study subjects will undergo a screening visit to assess eligibility after which a baseline metabolic assessment will be performed including a a fasting oral glucose tolerance test (OGTT) to measure normal glucose and insulin metabolism, an intravenous glucose tolerance test (IVGTT) to measure insulin sensitivity, MRI and DEXA scan to assess muscle and body fat distribution, VO2 max test and resting metabolic rate, and a muscle biopsy to look at how the muscle is affected by insulin and testosterone (T).

Subjects will then be randomized to one of three 12-week treatment arms, 1) Group 1 (Placebo); 2) Group 2 (Depot GnRH agonist (Zoladex) + Testosterone + placebo); or 3) Group 3 (Zoladex + Testosterone + aromatase inhibitor (anastrozole)). The rationale for this study design is as follows. Under normal physiological conditions, administration of T leads to a concomitant increase in estradiol (E2) levels due to endogenous conversion by the aromatase enzyme system. Therefore, in order to understand the relative roles of T and E2 on insulin sensitivity, one group of subjects will receive T in conjunction with the aromatase inhibitor, anastrozole.

At 13 weeks, the entire baseline evaluation including OGTT, IVGTT, resting metabolic rate and VO2 max, body composition assessment by DEXA and MRI, and muscle biopsy will be repeated. Subjects will return for a follow up visit four weeks later to measure CBC, T and PSA levels, to ensure levels are within the normal range.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 yr
* Diagnosis of the metabolic syndrome defined by the American Heart Association/National Heart, Lung, and Blood Institute guidelines as the presence of three or more of the following:

  * Waist circumference > 102 cm
  * Serum triglycerides > 150 mg/dL
  * HDL cholesterol < 40 mg/dL
  * Blood pressure > 130 mm Hg systolic or 85 mm Hg diastolic, or treatment with anti-hypertensives
  * Fasting serum glucose > 100 mg/dL
  * Plasma total testosterone level less than 300 ng/dL (1 SD below the mean for young healthy men)
  * Stable weight for previous three months (no weight change greater than or equal to +/-10 lbs)
  * Normal TSH, prolactin and prostate specific antigen (PSA) levels (<2.5 ng/mL)

Exclusion Criteria:

* New diagnosis of type 2 diabetes as defined by the ADA criteria: fasting glucose greater than 126 mg/dL or random blood glucose greater than 200 mg/dL on two occasions, or on oral hypoglycemic agents
* Contraindication to stress testing
* Contraindication to MRI scanning (Central nervous system aneurysm clips; Implanted neural stimulator; Implanted cardiac pacemaker or defibrillator; Cochlear implant; Ocular foreign body (e.g. metal shavings); Insulin pump; Metal shrapnel or bullet)
* History of testicular disorders (i.e. cryptorchidism)
* History of bleeding disorders (i.e. thrombocytopenia) or baseline hemoglobin levels less than 12g/dL
* History of metabolic bone disease (osteoporosis, osteomalacia)
* History of prostate cancer
* History of sleep apnea (subjects will also be excluded if at their baseline assessment they admit to heavy snoring, restless sleep, and/or excessive daytime somnolence)
* Symptoms of urinary outflow obstruction (i.e. benign prostatic hypertrophy)
* Illicit drug use or heavy alcohol use (>4 drinks/day)
* Allergic disorders
* Current medications (must exclude individuals taking the following medications):

  * Testosterone,
  * Cimetidine,
  * Spironolactone,
  * Ketoconazole,
  * Finasteride,
  * DHEA,
  * Androstenedione,
  * Oral steroids,
  * GnRH analogs

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2006-05; Primary Completion 2011-02 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
insulin sensitivity | at baseline and after 3 months

SECONDARY OUTCOMES:
glucose metabolism | at baseline and after 3 months
body composition VO2 max; resting metabolic rate; muscle biopsy analysis | at baseline and after 3 months
VO2 max | at baseline and after 3 months
resting metabolic rate | at baseline and after 3 months
muscle biopsy analysis | at baseline and after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Frances J Hayes, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Caronia LM, Dwyer AA, Hayden D, Amati F, Pitteloud N, Hayes FJ. Abrupt decrease in serum testosterone levels after an oral glucose load in men: implications for screening for hypogonadism. Clin Endocrinol (Oxf). 2013 Feb;78(2):291-6. doi: 10.1111/j.1365-2265.2012.04486.x. PMID 22804876